CLINICAL TRIAL: NCT00276614
Title: A Phase II Study of Bortezomib (Velcade ) Administered as a Single Agent in Metastatic Non-Clear Cell Renal Cell Carcinoma (RCC) Patients
Brief Title: Bortezomib in Treating Patients With Metastatic Kidney Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Jonsson Comprehensive Cancer Center (Other)
Collaborators: Millennium Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CDR0000453541; UCLA-0412011-01; MILLENNIUM-X05145
Record Dates: First submitted 2006-01-12; First posted 2006-01-13 (Estimated); Results first posted 2012-04-19 (Estimated); Last update posted 2020-09-01 (Actual); Status verified 2012-07

CONDITIONS: Kidney Cancer
Keywords: stage IV renal cell cancer; recurrent renal cell cancer; papillary renal cell carcinoma
MeSH Terms: conditions — Kidney Neoplasms; Carcinoma, Renal Cell | interventions — Bortezomib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Velcade (Experimental): Velcade IV twice a week for two weeks on Days 1, 4, 8 and 11 of each cycle. A 10 day-rest period (Days 12-21) with no Velcade will follow the 2 weeks of treatment in each cycle. one cycle = 21 days
  Interventions: Drug: bortezomib

INTERVENTIONS:
Drug: bortezomib

SUMMARY:
RATIONALE: Bortezomib may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth and by blocking blood flow to the tumor.

PURPOSE: This phase II trial is studying how well bortezomib works in treating patients with metastatic kidney cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Determine, preliminarily, the efficacy of bortezomib in patients with metastatic non-clear cell renal cell carcinoma in terms of objective response rate after a minimum of 2 courses of treatment.

Secondary

* Correlate clinical response in these patients with baseline von Hippel-Lindau expression and nuclear factor-KB activity.

OUTLINE: This is an open-label study.

Patients receive bortezomib IV over 3-5 seconds on days 1, 4, 8, and 11. Treatment repeats every 21 days for up to 6 courses in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed at 1 month and then periodically for 2 years.

PROJECTED ACCRUAL: A total of 27 patients will be accrued for this study.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed pure non-clear cell renal cell carcinoma (RCC)
* Distant metastatic disease (Tx, Nx, M1)
* Tumor expresses wild-type von Hippel-Lindau tumor suppressor gene/protein
* Measurable disease on imaging scan (≥ 1 cm)
* Brain metastases allowed provided they have been treated with surgery and/or radiation therapy and show no evidence of progression on cerebral CT or MRI scan 2 months following surgery and/or radiation therapy.
* Life expectancy ≥ 3 months
* Karnofsky performance status ≥ 60%
* Negative pregnancy test
* Fertile patients must use an acceptable method of contraception
* No other major illnesses likely to limit survival
* Platelet count ≥ 100,000/mm^3
* Absolute neutrophil count ≥ 1, 000/mm^3
* Hemoglobin ≥ 10 g/dL (transfusion allowed)
* Creatinine clearance ≥ 30 mL/min OR creatinine ≤ 2 mg/dL
* ALT or AST ≤ 2.5 times upper limit of normal
* At least 4 weeks since prior radiotherapy and recovered
* More than 30 days since any other prior investigational drugs

Exclusion Criteria:

* active CNS metastases
* pregnant or nursing
* myocardial infarction within the past 6 months
* New York Heart Association class III or IV heart failure
* uncontrolled angina
* severe uncontrolled ventricular arrhythmias
* electrocardiographic evidence of acute ischemia or active conduction system abnormalities
* Peripheral neuropathy ≤ grade 1
* hypersensitivity to bortezomib, boron, or mannitol
* history of a non-RCC malignancy within the past 5 years except basal cell carcinoma of the skin
* serious medical or psychiatric illness that would preclude study participation
* prior cytotoxic chemotherapy for this cancer
* other concurrent investigational therapy
* concurrent chemotherapy, immunotherapy, or hormonal therapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2006-04; Primary Completion 2009-07 (Actual); Study Completion 2009-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Matthew B. Rettig, MD, Study Chair — Jonsson Comprehensive Cancer Center
Locations (1):
- Jonsson Comprehensive Cancer Center at UCLA, Los Angeles, California, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment period from April 2006 through May 2009 at outpatient oncology clinic.
Groups:
- Bortezomib: Bortezomib 1.3 mg/m2 given on days 1, 4, 8, 11 of a 21 day cycle.
Period: Overall Study
Arm/Group | Bortezomib
Started | 4
Completed | 1
Not Completed | 3
Not completed — Progression of disease under study | 3

BASELINE CHARACTERISTICS:
Arm/Group | Bortezomib
Number analyzed (Participants) | 4
Age, Continuous [Median (Full Range); unit: years] | 42 [26 to 63]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1
  Male | 3
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 4
  More than one race | 0
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: Objective Response Rate as Measured by RECIST Criteria After Every 2 Courses of Treatment for up to 6 Courses
Time Frame: 2 months
Population: 2 subjects were excluded from analysis as they completed less than 2 cycles of study therapy.
Measure: Number; unit: participants
Arm/Group | Bortezomib
Number analyzed (Participants) | 2
participants | 2

ADVERSE EVENTS:
Time Frame: Beginning of treatment through 30 days post last treatment.
Arm/Group | Bortezomib
Serious Adverse Events (participants affected / at risk) | 0/4
Other Adverse Events (participants affected / at risk) | 2/4
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Bortezomib (N=4)
Thrombocytopenia (Blood and lymphatic system disorders) | 1 (1)
Nausea (Gastrointestinal disorders) | 1 (1)
Vomiting (Gastrointestinal disorders) | 1 (1)

LIMITATIONS AND CAVEATS:
Approval of several agents for management of renal cell carcinoma rendered accrual to this trial quite difficult.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No